CLINICAL TRIAL: NCT00418301
Title: Changes in Regional Cerebral Blood Flow as an Indicator of Neuronal Activity in Patients Treated With Spinal Cord Stimulation for Low Back and Leg Pain
Brief Title: Changes in Cerebral Blood Flow in Patients Treated With Spinal Cord Stimulation for Low Back and Leg Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCS0305
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Results first posted 2021-06-18 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-05

CONDITIONS: Pain; Low Back Pain; Leg Pain
Keywords: Pain; Neurostimulation
MeSH Terms: conditions — Pain; Low Back Pain | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Precision Spinal Cord Stimulation and PET Scan (Experimental): Positron emission tomography (PET) scan imaging procedures to assess Spinal Cord Stimulation.
  Interventions: Other: Precision Spinal Cord Stimulation and PET Scan

INTERVENTIONS:
Other: Precision Spinal Cord Stimulation and PET Scan — Imaging procedure to assess spinal Cord Stimulation.

SUMMARY:
The primary objective of this study is to identify the brain regions in which activity is affected by SCS. Baseline cerebral blood flow scans with the device turned off will be generated compared to scans produced with the device operating at parameters which produce optimal coverage of the painful areas. The relationship between cerebral blood flow and pain rating scores will be evaluated in both conditions.

DETAILED DESCRIPTION:
Spinal Cord Stimulation (SCS) is known to be effective in pain management. Some evidence exists that SCS may cause changes in cerebral blood flow. This study will be a novel PET examination of activity in brain regions affected by SCS. This activity will be compared with the pain intensity and distribution. Further, by examining cerebral blood flow at different doses of stimulation, relationships between SCS, brain perfusion, and pain relief can be drawn. This study will contribute to the elucidation of the mechanism of action of SCS.

ELIGIBILITY:
Inclusion Criteria:

* Have had one or more back surgery procedures.
* Have used an active Precision SCS device for chronic low back and bilateral leg pain for at least 6 weeks.
* Have bilateral leg pain.
* Have a baseline VAS of >4 (without stimulation).
* Have greater than 50% reduction in pain with SCS at optimal settings
* Be 18 years of age or older.
* Have the cognitive and functional capability to operate the controls for the device, to comply with directions during the study, and willing to participate in all study activities.
* Be capable of reading and understanding patient information materials and giving written informed consent.

Exclusion Criteria:

* Have any significant medical condition that is likely to interfere with study procedures or likely to confound evaluation of study endpoints.
* Have undergone a surgical lead revision or had any Precision components replaced after initial implantation.
* Are allergic to any of the injected media.
* Are pregnant or lactating.
* Have any contraindication to the PET scan procedure itself or exposure to the intravenous radioactive tracer (H215O).
* Have participated in any drug or device trial in the last 4 weeks or are currently participating in another drug or device trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Rauck, MD, Principal Investigator — Center for Clinical Research
Locations (1):
- Center for Clinical Research, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Precision Spinal Cord Stimulation and PET Scan
Started | 15
Completed | 12
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Efforts were made but the information is not accessible at this time. Hence baseline measures are not reported.
Arm/Group | Precision Spinal Cord Stimulation and PET Scan
Number analyzed (Participants) | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Cerebral Blood Flow and VAS With Optimal Paresthesia Coverage Compared With SCS Off
Time Frame: Within a few hours
Population: Efforts were made but the information is not accessible at this time. Hence outcome measures are not reported.
Arm/Group | Precision Spinal Cord Stimulation and PET Scan
Number analyzed (Participants) | 0

2. Secondary Outcome: Cerebral Blood Flow and VAS With Partial Paresthesia Coverage and Subthreshold Stimulation Compared With Optimal Coverage and With SCS Off
Time Frame: Within a few hours
Population: Efforts were made but the information is not accessible at this time. Hence outcome measures are not reported.
Arm/Group | Precision Spinal Cord Stimulation and PET Scan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment through end of study.
Description: Efforts were made but the information is not accessible at this time. Hence adverse events not reported.
Arm/Group | Precision Spinal Cord Stimulation and PET Scan
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes